CLINICAL TRIAL: NCT00058526
Title: A Multicenter Phase I Open-label Dose-escalation Vaccine Trial of dHER2 Protein With AS15 Adjuvant in HER2-overexpressing Patients With High-risk Breast Cancer
Brief Title: A Dose-escalation Vaccine Trial in HER2-overexpressing Patients With High-risk Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 719125/002; 104482 (Other: GlaxoSmithKline)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms, Breast
Keywords: dHER2-AS15 ASCI; Immunotherapeutic; Dose escalation; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (4):
- Cohort 1 (Experimental): Six doses of dHER2 (20 µg) + AS15 administered at Weeks 0, 2, 4, 6, 10 and 14.
  Interventions: Biological: Immunotherapeutic SB719125 (Primary)
- Cohort 2 (Experimental): Six doses of dHER2 (100 µg) + AS15 administered at Weeks 0, 2, 4, 6, 10 and 14.
  Interventions: Biological: Immunotherapeutic SB719125 (Primary)
- Cohort 3 (Experimental): Six doses of dHER2 (500 µg) + AS15 administered at Weeks 0, 2, 4, 6, 10 and 14. Patients in this cohort can receive two booster doses at Weeks 34 and 38, respectively.
  Interventions: Biological: Immunotherapeutic SB719125 (Primary)
- Cohort 4 (Experimental): Three doses of dHER2 (20 µg) + AS15 administered at Weeks 0, 4, and 14. Patients in this cohort can receive two booster doses at Weeks 34 and 38, respectively.
  Interventions: Biological: Immunotherapeutic SB719125 (Primary)

INTERVENTIONS:
Biological: Immunotherapeutic SB719125 (Primary) — Intramuscular injection
  Other Names: dHER2 ASCI

SUMMARY:
Treatment phase:

The purpose of this study is to evaluate the safety and the immune response elicited by a new anti-cancer therapy in patients with breast cancer in remission but who are at high risk of relapse. The study product is an immunotherapeutic consisting of the recombinant dHER2 protein combined with an immunostimulant called AS15. The study aims to determine the optimal of three different dose levels of dHER2 combined with the same fixed dose of AS15 by assessing the safety and the immune response elicited after a series of injections of the study product.

Five-year follow-up phase:

This part of the study aims to assess any late onset toxicity of the study treatment through yearly follow-up visits and to monitor the patients' survival and disease status up to five years after the last administration of the study treatment. The patients' immune response is also measured to assess the robustness of the immune response elicited by the study treatment.

ELIGIBILITY:
Inclusion criteria:

1. Patient must have a previous diagnosis of HER2/neu-positive breast cancer: FISH positive test (for HercepTest 2+ patients), or, HercepTest 3+ patients.
2. Patients must be Stage II with at least one positive node or Stage III in remission. Patients must have had standard treatment for their cancer, including lymph node dissection and at least one course of standard adjuvant treatment.
3. Patient must have completed at least one course of standard adjuvant treatment within 5 years of study entry.
4. Patient may be on concurrent hormonal therapy.
5. Patient must be free of recurrent breast cancer as shown by standard diagnostic tests at entry onto study.
6. Patient must have a chest X-ray showing no evidence of disease.
7. Patient should have an expected survival of at least 12 months.
8. Written informed consent must be obtained prior to any protocol-specific procedures being performed.
9. Patient must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0.
10. Patient must not be pregnant and must use adequate contraception throughout the study and must plan to not bear children in the future.
11. Patient must not be lactating.
12. Patient must have a negative pregnancy test prior to enrollment. Pregnancy testing need not be done for patients who are > 55 years of age, post-menopausal or surgically sterile.
13. Patient must be 40 to 70 years of age inclusive. Patients younger than 40 years of age may be enrolled if they are sterile and incapable of childbearing. Chemotherapy-induced amenorrhea is not considered to be a sign of sterility.
14. Patient must have adequate bone marrow reserve as indicated by: WBC ≥3000/mm3, neutrophils ≥1500/ mm3, platelets ≥100,000 mm3, lymphocytes ≥1000/mm3, and hemoglobin ≥10.0 g/dL.
15. Patient must have an absolute CD4 cell count of >200 cells/mm3.
16. Patient must have adequate renal function.
17. Patient must have adequate hepatic function as indicated by: serum bilirubin within normal limits, aspartate aminotransferase <1.5 times the upper limit of normal and an alkaline phosphatase <1.2 times the upper limit of normal. Patients with an alkaline phosphatase above normal must have negative bone scans and abdominal CT scans prior to entry onto protocol.
18. Patient must have a baseline left ventricular ejection fraction (LVEF) measured by multi-gated acquisition (MUGA) scan equal to or greater than the lower limit of normal for the radiology facility. The serial MUGA scans for each individual must also be performed at the same radiology facility, using the same equipment in the same manner, for consistency of method.
19. Patients who had an earlier baseline MUGA scan at the radiological facility of the investigator's site to be used in the study, such as a MUGA scan done prior to adjuvant treatment, must meet the above criteria for LVEF AND must also not have had a decrease in LVEF of above 15 percentage points from the original baseline MUGA scan. Patients who have not had a MUGA scan done at this radiological facility prior to adjuvant treatment must have a normal MUGA scan at screening.
20. Patient must not be known to be HIV positive. Results of virology screening must indicate that the patient has negative serology for HCV (hepatitis C virus) and is negative for HBsAg (hepatitis B surface antigen). (HBV testing indicating positive serology (antibodies) is allowed.)

Exclusion criteria:

1. Patients who are presently being treated with Herceptin or have been treated with Herceptin in the past.
2. Patients who have received surgery or chemotherapy treatments within 8 weeks prior to enrollment. Patients who have received radiation therapy within 12 weeks prior to enrollment.
3. Patients who have received > 300 mg/m2 doxorubicin (cumulative dose) or > 600 mg/m2 epirubicin (cumulative dose).
4. Patients with any uncontrolled bleeding disorder or coagulation disorder or thrombocytopenia or prothrombotic disorder.
5. Patients with auto-immune disease such as, but not limited to multiple sclerosis, lupus, and inflammatory bowel disease, Graves' disease and Hashimoto's disease.
6. Patients with a history of previous anaphylaxis or severe allergic reaction to vaccines or unknown allergens.
7. Patients with previous splenectomy or radiation to the spleen.
8. Patients who have received a major organ graft (including bone-marrow transplantation).
9. Patients who require chronic oral treatment (defined as more than 14 days) with immunosuppressive agents including glucocorticosteroids or other immune-modifying drugs.
10. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for > 2 years and highly likely to have been cured.
11. Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to unacceptable risk.
12. Patients with previous congestive heart failure or difficult-to-control hypertension. Patients with known coronary artery disease, arrhythmia requiring treatment, clinically significant valvular disease, cardiomegaly on chest X-ray, ventricular hypertrophy on electrocardiogram (EKG) or previous myocardial infarction.
13. Patients with psychiatric or addictive disorders that may compromise the ability to give informed consent, or comply with the trial procedures.
14. Patients who have received any investigational or non-registered drug or non-registered vaccine other than the study product within the 30 days preceding the first dose of study product, or who plan to receive such a drug during the study period.
15. Patients who have received any immunoglobulins and/or blood products within the 3 weeks prior to study product administration.
16. Patients who have received any commercial vaccine within one week before the first dose of the study product.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-03-20 (Actual); Primary Completion 2006-09-06 (Actual); Study Completion 2006-09-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity (DLT) | During the study period (until Week 40 or 43) and the post-study follow-up period (5 years)
Occurrence of cardiotoxicity | During the study period (until Week 40 or 43) and the post-study follow-up period (5 years)
Occurrence of Grade 3 or 4 adverse events | During the study period (until Week 40 or 43) and the post-study follow-up period (5 years)
Occurrence of solicited local and general signs and symptoms recorded by the patient on diary cards | Period of eight days (Day 0 to Day 7) immediately after each administration of the study treatment
Occurrence of unsolicited non-serious adverse events | During the study period (until Week 40 or 43) and the post-study follow-up period (5 years)
Occurrence of serious adverse events | During the study period (until Week 40 or 43) and the post-study follow-up period (5 years)
Hematological, biochemical (including auto-immunity) and urinalysis parameters | During the study period (until Week 40 or 43)
Changes in vital signs | During the entire study period (until Week 40 or 43)
Physical examination findings | During the study period (until Week 40 or 43)

SECONDARY OUTCOMES:
Anti-dHER2, anti-HER2 ECD (extracellular domain), anti-HER2 ICD (intracellular domain) antibody concentrations | Two weeks after the fourth and sixth study treatment administrations (Week 6 and Week 14) and at the three and six months follow-up visit (Week 26 and Week 40). At yearly visits during the five-year follow-up period
Anti-dHER2, anti-HER2 ECD and anti-HER2 ICD seropositivity | Two weeks after the fourth and sixth study treatment administrations (Week 6 and Week 14) and at the three and six months follow-up visit (Week 26 and Week 40). At yearly visits during the five-year follow-up period
In vitro functional activity response (e.g. growth inhibition of HER2-overexpressing breast tumor cells) expressed as a percentage of inhibition | After four or six administrations of the study treatment
Antibody-dependent cellular cytotoxicity (ADCC, % of lysis) - optionally | After four or six administrations of the study treatment
In vitro cellular immune response to dHER2, HER2 ECD and HER2 ICD as shown by lymphoproliferative response (expressed by stimulation index) and by secretion of interferon-γ and interleukin-5 expressed by concentration (pg/mL) | At baseline, after Dose 4, after Dose 6, at six months follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (4):
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Seattle, Washington
- Australia (3):
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Leuven
- France (3):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Herblain
- Italy (3):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Perugia, Umbria

REFERENCES:
- [Derived] Limentani SA, Campone M, Dorval T, Curigliano G, de Boer R, Vogel C, White S, Bachelot T, Canon JL, Disis M, Awada A, Berliere M, Amant F, Levine E, Burny W, Callegaro A, de Sousa Alves PM, Louahed J, Brichard V, Lehmann FF. A non-randomized dose-escalation Phase I trial of a protein-based immunotherapeutic for the treatment of breast cancer patients with HER2-overexpressing tumors. Breast Cancer Res Treat. 2016 Apr;156(2):319-30. doi: 10.1007/s10549-016-3751-x. Epub 2016 Mar 18. PMID 26993131
- See also: Results for study 719125/002 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/719125/002?search=study&#rs